CLINICAL TRIAL: NCT04998773
Title: Efficacy, Clinical and Neuroimaging Biomarkers of Response of Two Intensive/Spaced Protocols of Theta-Burst Transcranial Magnetic Stimulation in Resistant Depression: a Randomized Double-blinded Placebo-controlled Clinical Trial
Brief Title: Efficacy and Biomarkers of Response of TBS in Treatment Resistant Depression
Acronym: EMTtfNI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Spanish Agency of Medicines and Health Products (Other Government); Hospital Universitario La Fe (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Pilar Sierra Sanmiguel, Principal Investigator, Leader of Mental Health Investigation Group, Instituto de Investigacion Sanitaria La Fe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-326-1; PI 2022-280-1 (Other Grant/Funding Number: Carlos III Health Institute); 21-0040 (Other: AEMPS, NEOPS code)
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Resistant Depression, Treatment; Bipolar Depression
Keywords: TMS; iTBS; Depression; Bipolar depression; Antidepressants; Neuroimaging; PET-MRI
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group Bilateral (Active Comparator): 32 patients, bilateral active TBS stimulation, Will receive an intensive-spaced protocol Intermittent TBS in left DLPFC and Continuous TBS in right DLPFC
  Interventions: Device: Theta Burst Transcranial Magnetic Bilateral Stimulation
- Group Unilateral (Active Comparator): 32 patients, unilateral left DLPFC active TBS stimulation. Will receive an intensive-spaced protocol Intermittent TBS in left DLPFC and Sham Continuous TBS in right DLPFC
  Interventions: Device: Theta Burst Transcranial Magnetic Unilateral Stimulation
- Group Placebo (Placebo Comparator): 32 patients, bilateral sham TBS stimulation. Will receive an intensive-spaced protocol of Sham Intermittent TBS in left DLPFC and Sham Continuous TBS in right DLPFC
  Interventions: Device: Theta Burst Transcranial Magnetic Sham Stimulation

INTERVENTIONS:
Device: Theta Burst Transcranial Magnetic Bilateral Stimulation — TMS protocol of 22 sessions of bilateral active 1800 pulses.
  Arms: Group Bilateral
Device: Theta Burst Transcranial Magnetic Sham Stimulation — TMS protocol of 22 sessions of sham bilateral 1800 pulses.
  Arms: Group Placebo
Device: Theta Burst Transcranial Magnetic Unilateral Stimulation — TMS protocol of 22 sessions of left active 1800 pulses and right sham 1800 pulses.
  Arms: Group Unilateral

SUMMARY:
Theta Burst Transcranial Magnetic Stimulation (TBS) in dorsolateral prefrontal cortex (DLPFC) has shown efficacy and safety as an adjuvant strategy for resistant to treatment depression (RTD) in daily sessions during 4-6 weeks (20-30 sessions). Current investigation in TBS aims to design intensive treatment protocols so as to achieve earlier responses and higher rates of efficacy. However, the implementation of TBS in the Public National Health Service requires cost-effective protocols that ensure and facilitate patients adherence to treatment, and whose design is based on clinical and neuroimaging biomarkers of response so as to adequately select candidate patients. The aim of this study is to assess the efficacy and safety of novel bilateral and unilateral intensive and spaced protocols of TBS in outpatients with unipolar and bipolar RTD compared with sham stimulation. Specific objectives: I) Comparison of mood change, response and remission of depressive illness at the end of TBS protocol in the groups and maintenance of its effect at 3 months; II) Characterization of neuroimaging cerebral connectivity networks and cerebral metabolism patterns of patients with RTD related to the effects of bilateral or unilateral TBS; III) Identification of clinical and demographic predictors contributing to response to TBS; IV) Analysis of the interaction between clinical, demographic and neuroimaging predictors so as to determine a RTD profile of patient that can benefit from TBS.

DETAILED DESCRIPTION:
Participants will receive 22 bilateral sessions of sham/active continuous (right DLPFC) and intermittent (left DLPFC) TBS during 6 weeks. Simultaneous cerebral PET-MRI will be performed before (week 0) and after the treatment with TBS (week 7)

* Weeks 1 and 2: 1 session 5 days a week (10 sessions)
* Weeks 3,4,5, 6: 1 session 3 days a week (12 sessions)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Episode or Depressive phase in Bipolar Disorder DSM-5 criteria.
* Moderate severity (>14 points in HDRS)
* 2 antidepressant failures or failure in enhancing strategies in the case of bipolar depression.
* No changes in treatment 3 week previous to the onset of treatment with TMS.
* Ability to sign informed consent.

Exclusion Criteria:

* Any psychiatric comorbidity in axis I or II.
* Depressive episode with psychotic features.
* Dysthymia.
* Treatment with ECT in current depressive episode.
* Multiresistance (> 6 trials of therapeutic strategies).
* Suicide risk assessed previous to each session.
* Patients who miss 2 TMS sessions in a row
* Neurological comorbidities (epilepsy, Parkinson disease, neurocognitive disorders).
* Contraindications to TMS: pregnancy, metallic cervical or head implants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale 17 items (HDRS-17) at the end of the treatment respect to basal. | 6 weeks
  Hetero-administered

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II) respect to basal. | 2, 6 weeks
  Self-administered
Montgomery Asberg Depression Rating Scale (MADRS) respect to basal. | 2, 6 weeks
  Hetero-administered
Young Mania Rating Scale (YMRS) at the end of the treatment respect to basal. | 2, 6 weeks
  Hetero-administered
Altman Self Rating Mania Scale (ASRM) at the end of the treatment respect to basal. | 2, 6 weeks
  Self-administered
Clinical Global Impression Scale (CGI) respect to basal. | 2,6 weeks
  Hetero-administered
Hamilton Anxiety Scale (HAM-A) respect to basal. | 2,6 weeks
  Hetero-administered
Oviedo Sleep Questionnaire (OSQ) respect to basal. | 2, 6 weeks
  Hetero-administered
Dimensional Apathy Scale (DAS) respect to basal | 6 weeks
  Self-administered
Screening for Cognitive Impairment por Psychiatry (SCIP) at the end of the treatment respect to basal. | 6 weeks
  Hetero-administered (versions A and B)
Short Form Health Survey (SF 36) at the end of the treatment respect to basal. | 6 weeks
  Self-administered
Functional Assessment Short Test (FAST) at the end of the treatment respect to basal. | 6 weeks
  Hetero-administered
Global assessment of Functioning (GAF) at the end of the treatment respect to basal. | 6 weeks
  Hetero-administered
Response to treatment | 2 and 6 weeks
  50% reduction in HDRS-17
Response to treatment | 2 and 6 weeks
  50% reduction in MADRS
Remission | 2 and 6 weeks
  HDRS-17<8 points
Remission | 2 and 6 weeks
  MADRS<11 POINTS

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Sierra San Miguel, PhD, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Fitzgerald PB, Chen L, Richardson K, Daskalakis ZJ, Hoy KE. A pilot investigation of an intensive theta burst stimulation protocol for patients with treatment resistant depression. Brain Stimul. 2020 Jan-Feb;13(1):137-144. doi: 10.1016/j.brs.2019.08.013. Epub 2019 Aug 22. PMID 31477542
- [Background] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188